CLINICAL TRIAL: NCT03995264
Title: Ultrasound vs Palpation for Radial Artery Cannulation in Patients Undergoing Bariatic Surgery
Brief Title: Ultrasound vs Palpation for Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJIRB-MED-THE-19-148
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Ultrasound-guided radial artery cannulation
  Interventions: Procedure: Ultrasound -guided cannulation
- Palpation group (Placebo Comparator): Radial artery cannulation with palpation technique
  Interventions: Procedure: Palpation -guided cannulation

INTERVENTIONS:
Procedure: Ultrasound -guided cannulation — radial artery cannulation using the ultrasound
  Arms: Ultrasound group
Procedure: Palpation -guided cannulation — radial artery cannulation using the palpation
  Arms: Palpation group

SUMMARY:
The primary purpose of this study is to compare the palpation technique with ultrasound guidance for radial artery cannulation for bariatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists 1, 2, 3 BMI ≥ 30 bariatic surgery

Exclusion Criteria:

* refusal infection or surgery history in wrist

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Success rate | at first attempt, as average 5 min
  Success rate at first attempt for radial artery cannulation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoul, South Korea

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140